CLINICAL TRIAL: NCT06304311
Title: Effectiveness of Backside Massage and Lamaze Breathing on Labour Outcome Among Primigravida in Tertiary Care Hospitals, Lahore Pakistan: A Randomized Control Trial
Brief Title: Effectiveness of Backside Massage and Lamaze Breathing on Labour Outcome Among Primigravida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Collaborators: Mahsa University (Other)
Responsible Party: Principal Investigator, Muhammad Mansoor Hafeez, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MAHSA/PHD/SON/2024/01
Record Dates: First submitted 2024-02-11; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Obstetrics care (Control) (Active Comparator): Participants in the control arm received routine obstetrics care, which typically includes standard prenatal care, monitoring during labor, and delivery management according to established hospital protocols. There were no additional interventions or techniques implemented beyond standard practice for managing labor and delivery.
  Interventions: Procedure: Routine Obstetrics care & Lamaze breathing techniques and backside massage
- Routine Obstetrics care & Lamaze breathing techniques and backside massage (Interventional group) (Experimental): Participants in the experimental arm received routine obstetrics care, similar to the control group, along with additional interventions of Lamaze breathing techniques and backside massage. Lamaze breathing techniques were taught to participants during antenatal classes or individual sessions, focusing on deep breathing, relaxation, and pain management strategies during labor. Backside massage was administered by trained personnel using gentle, rhythmic strokes on the lower back to alleviate discomfort and promote relaxation during labor. These interventions were integrated into the labor and delivery process alongside routine obstetrics care.
  Interventions: Procedure: Routine Obstetrics care & Lamaze breathing techniques and backside massage

INTERVENTIONS:
Procedure: Routine Obstetrics care & Lamaze breathing techniques and backside massage — Lamaze breathing techniques Five breathing patterns were introduced namely- cleansing breathing for relaxation, slow-paced breathing, modified-paced breathing and patterned- paced breathing. These patterns were used during and following contractions. Gentle pushing, and breath-hold during pushing were instructed during the second stage of labor which encouraged descent of the baby.
  Backside massage during 2nd stage of labor by the trained massage therapist.

SUMMARY:
The study aims to investigate the effects of a combination of Lamaze breathing exercises and backside massage on the labor experiences of primigravidae in Pakistan. Labour pain, if left unaddressed, can lead to abnormal labor, hence the importance of effective pain management techniques. Lamaze breathing techniques are non-pharmacological methods aimed at psychologically and physically preparing mothers for drug-free childbirth. Backside massage therapy is another non-invasive intervention that can help to reduce pain and anxiety during labor. The study will involve a randomized controlled trial with two groups: an intervention group receiving backside massage and Lamaze breathing along with standard labor care, and a control group receiving only standard labor care. Primigravidae between 26 to 34 weeks of gestation without chronic diseases or pregnancy-related complications will be recruited from antenatal departments. Eligible participants will be randomly allocated to either group to minimize bias. The backside massage therapy intervention will be administered by trained massage therapists. Outcome measures include level of labor pain and anxiety levels, maternal stress hormone levels (adrenocorticotropic hormone, cortisol, and oxytocin), maternal vital signs, fetal heart rate, labor duration, APGAR scores, and maternal satisfaction and self-efficacy. The sample size of 90 participants (45 in each group) has been determined to achieve a 95% power level with a 5% error rate, accounting for a 20% attrition rate. Data analysis will employ mixed-effect regression models, time series analyses, paired t-tests, or equivalent non-parametric tests to assess between-group and within-group outcome measures. The study aims to provide valuable insights into the efficacy of combining Lamaze breathing exercises and backside massage therapy as complementary interventions for managing labor pain and anxiety among primigravidae in Pakistan, potentially reducing the need for medically unnecessary cesarean sections and improving maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primigravidae
* Age 20-35 years old
* Gestational age of 37-41 weeks
* First stage of labour
* Singleton pregnancy
* Cephalic presentation
* Regular contractions
* Cervical dilatation of at least 6 cm
* Minimum of three contractions every 10 minutes
* Contraction intensity of at least moderate
* Contraction duration between 30 seconds and 60 seconds

Exclusion Criteria:

* Diagnosis of underlying chronic diseases (e.g., cardiovascular disease, kidney disease, diabetes, asthma, mental health disorders, epilepsy or seizure)
* Pregnancy-related diseases (e.g., gestational diabetes, preeclampsia, cephalo-pelvic disproportion, polyhydramnios or oligohydramnios, deep venous thrombosis)
* Pregnancy complications (e.g., placenta praevia, antepartum haemorrhage, fetal distress, administration of analgesics)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Labour pain intensity | During 1st stage to 01 day after labour
  Labour pain intensity is a measure used to assess the severity or level of pain experienced by a woman during childbirth. It typically involves asking the woman to rate her pain on a scale, often ranging from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable. This outcome measure helps healthcare providers understand the woman's level of discomfort during Labour and can guide decisions regarding pain management strategies and interventions to ensure her comfort and well-being throughout the birthing process.
Anxiety level | During 1st stage to 01 day after labour
  Anxiety levels were measured by GAD-7 scoring system. GAD-7 is a brief self-report questionnaire designed to screen for generalized anxiety disorder and assess its severity. It consists of 7 items, and participants rate how often they have been bothered by each symptom over the past two weeks on a scale from 0 to 3. Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Duration of Labour | During 1st stage to 01 day after labour
  Duration of labour is a measure used to assess the length of time it takes for a woman to progress through the stages of childbirth, from the onset of regular contractions to the delivery of the baby and placenta. It is typically recorded in hours or minutes and includes the duration of both the active and passive phases of labour, as well as the length of time spent pushing during the second stage. Monitoring the duration of labour is essential for healthcare providers to evaluate the progress of labour, identify potential complications, and make informed decisions regarding interventions or assistance to ensure a safe and healthy delivery for both the mother and baby.
Maternal self-efficacy | During 1st stage to 01 day after labour
  Childbirth Self-Efficacy Inventory (CBSEI) for the measurement of maternal confidence & self-efficacy By Nancy. K. Lowe, for the experimental and control group. (Tool indicates 1 which indicates not all helpful and 10 very helpful)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Lim Gek Mul, Study Chair — Masha University; Prof. Dr. Rusli Bin Nordin, Study Director — Masha University
Locations (1):
- Lady Wallingdon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Till the publication of data nothing will be share